CLINICAL TRIAL: NCT03283904
Title: Active Schools: Skelmersdale
Acronym: AS:Sk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edge Hill University (Other)
Collaborators: West Lancashire Sport Partnership (Unknown); West Lancashire Leisure Trust (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KIDSMOVE
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Physical Activity; Sedentary Lifestyle
Keywords: Children; Schools
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Control vs Intervention clusters of schools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multicomponent PA intervention (Experimental): Intervention schools will adopt a multicomponent intervention by integrating physical activities into different parts of the school day
  Interventions: Other: Multicomponent physical activity intervention

INTERVENTIONS:
Other: Multicomponent physical activity intervention — School-based multicomponent intervention

SUMMARY:
The aim of AS:Sk is to improve physical activity levels and health-related outcomes of children from the Skelmersdale area of West Lancashire through a school-based physical activity multi-component intervention.

DETAILED DESCRIPTION:
The multi-component intervention is the third and final phase of the AS:Sk project. It will be implemented and evaluated in four of the seven participating schools. The remaining three schools will act as controls and will not implement any physical activity intervention during the period of the research project. Schools will be randomly assigned to either intervention or control conditions. The multi-component intervention will involve multiple areas of the schools' curricula, environments, or policies being targeted. Decisions regarding these intervention components will be influenced by what was deemed effective, and feasible within phase 2 of the project. Phase 2 included a four week trial of three different single component physical activity interventions across all participating schools. Phase 3 will be implemented for at least eight weeks and if successful, it would then be rolled out in the control schools at the end of the project. Participants from both intervention and control schools will take part in the measures for evaluation in this third and final phase of the project.

ELIGIBILITY:
Inclusion Criteria:

* Year 5 pupil attending participating schools

Exclusion Criteria:

-

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
School-day moderate-to-vigorous physical activity (MVPA) | 7 days
  Minutes of school-day MVPA accrued

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Fairclough, Principal Investigator — Edge Hill University
Locations (1):
- Edge Hill University, Ormskirk, Lancs, United Kingdom

REFERENCES:
- [Result] Taylor SL, Curry WB, Knowles ZR, Noonan RJ, McGrane B, Fairclough SJ. Predictors of Segmented School Day Physical Activity and Sedentary Time in Children from a Northwest England Low-Income Community. Int J Environ Res Public Health. 2017 May 16;14(5):534. doi: 10.3390/ijerph14050534. PMID 28509887
- [Result] Fairclough SJ, Dumuid D, Taylor S, Curry W, McGrane B, Stratton G, Maher C, Olds T. Fitness, fatness and the reallocation of time between children's daily movement behaviours: an analysis of compositional data. Int J Behav Nutr Phys Act. 2017 May 10;14(1):64. doi: 10.1186/s12966-017-0521-z. PMID 28486972